CLINICAL TRIAL: NCT02346110
Title: Comparison of the Effect of a Single Shot Saphenous Block With Plain Bupivacaine vs. Protracted Bupivacaine Mixture as a Supplement to Continuous Sciatic Catheter After Major Ankle and Foot Surgery
Brief Title: Protracted Effect of the Ultrasound-guided Saphenous Block
Acronym: PEUSB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProtokolSB1; 2014-004207-78 (EudraCT Number)
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2015-10

CONDITIONS: Arthrosis, Unspecified, Ankle and Foot
MeSH Terms: conditions — Osteoarthritis | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine-adrenalin + sodium chloride (Active Comparator): Single shot saphenous block:
  10 mL of 5 mg/mL bupivacaine with 5 μg/mL adrenalin = 50 mg bupivacain and 50 μg adrenalin
  1 mL sodium chloride solution
  Interventions: Drug: Bupivacaine-adrenaline; Other: Sodium chloride
- Bupivacaine-adrenaline + Dexamethasone (Experimental): Single shot saphenous block:
  10 mL of 5 mg/mL bupivacaine with 5 μg/mL adrenalin = 50 mg bupivacain and 50 μg adrenalin
  1 mL of 4 mg/mL dexamethasone = 4 mg dexamethasone
  Interventions: Drug: Bupivacaine-adrenaline; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine-adrenaline — 50 mg bupivacaine and 50 μg adrenalin
  Other Names: Marcain-adrenalin
Drug: Dexamethasone — 4 mg
  Other Names: Dexagalen
  Arms: Bupivacaine-adrenaline + Dexamethasone
Other: Sodium chloride — 1 mL of sodium chloride solution as placebo
  Other Names: NaCL
  Arms: Bupivacaine-adrenalin + sodium chloride

SUMMARY:
This study focuses on optimizing the postoperative pain treatment after major foot and ankle surgery by prolonging the duration of the ultrasound-guided saphenous block. The currently used single shot saphenous block only covers half of the pain intensive period from the saphenous territory, which results in a sharp, break-through pain requiring opioids. The hypothesis is that this protracted mixture will keep the patients free of pain without the use of opioids for the entire pain intensive period and thus increase rehabilitation and patients' satisfaction.

DETAILED DESCRIPTION:
Half of the patients will receive a single shot saphenous block with 10 mL bupivacaine-adrenalin and 1 mL of sodium chloride solution, while the other half will receive 10 mL of bupivacaine-adrenalin and 1 mL of dexamethasone.

The block is strictly a sensory block because it is a selective, sub-sartorial saphenous block at mid-thigh level without any anesthetic effect on the femoral nerve.

The adjuvant dexamethasone has increasingly become a subject of interest regarding a protracted effect, which has been shown in several studies. However, the precise mechanism of action remains speculative, and the results are contradictory regarding the discussion whether the effect is systemic or local. The effect may stem from decreased nociceptive C-fibre activity via a direct action on glucocorticoid receptors and inhibitory potassium channels. Another suggestion is a vasoconstrictive effect, which reduces the systemic uptake of local anaesthetics or a systemic anti-inflammatory effect.

Prolonging the effect of the single shot saphenous block by adding dexamethasone will reduce the need for opioids, which will reduce the risk of adverse effects like nausea, vomiting and respiratory depression. Furthermore, newer studies show that inadequate pain alleviation in the early postoperative period is a risk factor in developing chronic persistent pain.

ELIGIBILITY:
Inclusion Criteria:

* Elective ankle or hind foot surgery either: (1) total ankle arthroplasty, (2) ankle arthrodesis or (3) subtalar arthrodesis
* Age ≥ 18
* American Society of Anaesthesiology Classification I-III
* Informed consent both orally and in writing after the patient has fully understood the protocol and its limitations.

Exclusion Criteria:

* Communication problems or dementia
* Allergies to any medical product used in the study
* Neuropathy of the sciatic or femoral nerve prior to the operation
* Morbus Charcot-Marie-Tooth disease, diabetic neuropathy, peripheral vascular disease
* BMI > 35
* Pregnancy
* Daily use of opioids
* Coagulation disorders
* Infection at the site of injection or systemic infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Duration of the saphenous nerve block | 48 hours
  The duration is registered as the time until the first dose of morphine is taken, and when the pain score is above 3 and located to the frontal or medial side of the ankle. Morphine is administered intravenously by a patient controlled pump (PCA - Patient Controlled Analgesia)

SECONDARY OUTCOMES:
Cumulated opioid consumption | 48 hours
  Registered by the PCA pump
Pain score | Arrival at the Perioperative Section which will be within 30 minutes after surgery. Departure from the Perioperative Section which is expected to be on average 2 hours after surgery. 6, 12, 24, 30, 36, 42 and 48 hours after surgery
  NRS (numeric rating scale)
Pain localization | Arrival at the Perioperative Section which will be within 30 minutes after surgery. Departure from the Perioperative Section which is expected to be on average 2 hours after surgery. 6, 12, 24, 30, 36, 42 and 48 hours after surgery
  Lateral or medial side of the ankle
Test of sensory block | Arrival at the Perioperative Section which will be within 30 minutes after surgery. Departure from the Perioperative Section which is expected to be on average 2 hours after surgery. 6, 12, 24, 30, 36, 42 and 48 hours after surgery
  The sensory block of the peroneal nerve is tested on the dorsal side of the toes and the tibial nerve on the plantar side of the toes.
  The ankle and lower leg is covered in cast, and therefore the saphenous nerve is tested around the tibial tuberosity because this area is innervated by the infra-patellar nerve, which is a branch of the saphenous nerve

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fichtner Bendtsen, MD, phD, Principal Investigator — Department of Anesthesiology, Aarhus University Hospital
Locations (1):
- Department of Anesthesiology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clendenen SR, Whalen JL. Saphenous nerve innervation of the medial ankle. Local Reg Anesth. 2013 Mar 6;6:13-6. doi: 10.2147/LRA.S42603. Print 2013. PMID 23630434
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Blumenthal S, Borgeat A, Neudorfer C, Bertolini R, Espinosa N, Aguirre J. Additional femoral catheter in combination with popliteal catheter for analgesia after major ankle surgery. Br J Anaesth. 2011 Mar;106(3):387-93. doi: 10.1093/bja/aeq365. Epub 2010 Dec 17. PMID 21169609
- [Background] Cepeda MS, Farrar JT, Baumgarten M, Boston R, Carr DB, Strom BL. Side effects of opioids during short-term administration: effect of age, gender, and race. Clin Pharmacol Ther. 2003 Aug;74(2):102-12. doi: 10.1016/S0009-9236(03)00152-8. PMID 12891220
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Richman JM, Liu SS, Courpas G, Wong R, Rowlingson AJ, McGready J, Cohen SR, Wu CL. Does continuous peripheral nerve block provide superior pain control to opioids? A meta-analysis. Anesth Analg. 2006 Jan;102(1):248-57. doi: 10.1213/01.ANE.0000181289.09675.7D. PMID 16368838
- [Background] Ya Deau JT, Wukovits BU, LaSala VR, Jules-Elysee KM, Paroli L, Kahn RL, Levine DS, Lipnitsky JY. Similar analgesic effect after popliteal fossa nerve blockade with 0.375% and 0.75% bupivacaine. HSS J. 2007 Sep;3(2):173-6. doi: 10.1007/s11420-007-9052-5. PMID 18751790
- [Background] Borgeat A, Blumenthal S, Lambert M, Theodorou P, Vienne P. The feasibility and complications of the continuous popliteal nerve block: a 1001-case survey. Anesth Analg. 2006 Jul;103(1):229-33, table of contents. doi: 10.1213/01.ane.0000221462.87951.8d. PMID 16790658
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Bendtsen TF, Moriggl B, Chan V, Pedersen EM, Borglum J. Defining adductor canal block. Reg Anesth Pain Med. 2014 May-Jun;39(3):253-4. doi: 10.1097/AAP.0000000000000052. No abstract available. PMID 24747312
- [Background] Chen J, Lesser J, Hadzic A, Resta-Flarer F. The importance of the proximal saphenous nerve block for foot and ankle surgery. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):372. doi: 10.1097/AAP.0b013e318295596a. No abstract available. PMID 23788076
- [Background] Forster JG, Rosenberg PH. Clinically useful adjuvants in regional anaesthesia. Curr Opin Anaesthesiol. 2003 Oct;16(5):477-86. doi: 10.1097/00001503-200310000-00007. PMID 17021500
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Kawanishi R, Yamamoto K, Tobetto Y, Nomura K, Kato M, Go R, Tsutsumi YM, Tanaka K, Takeda Y. Perineural but not systemic low-dose dexamethasone prolongs the duration of interscalene block with ropivacaine: a prospective randomized trial. Local Reg Anesth. 2014 Apr 5;7:5-9. doi: 10.2147/LRA.S59158. eCollection 2014. PMID 24817819
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Rahangdale R, Kendall MC, McCarthy RJ, Tureanu L, Doty R Jr, Weingart A, De Oliveira GS Jr. The effects of perineural versus intravenous dexamethasone on sciatic nerve blockade outcomes: a randomized, double-blind, placebo-controlled study. Anesth Analg. 2014 May;118(5):1113-9. doi: 10.1213/ANE.0000000000000137. PMID 24686045
- [Background] Shrestha BR, Maharjan SK, Tabedar S. Supraclavicular brachial plexus block with and without dexamethasone - a comparative study. Kathmandu Univ Med J (KUMJ). 2003 Jul-Sep;1(3):158-60. PMID 16388222
- [Background] Parrington SJ, O'Donnell D, Chan VW, Brown-Shreves D, Subramanyam R, Qu M, Brull R. Dexamethasone added to mepivacaine prolongs the duration of analgesia after supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):422-6. doi: 10.1097/AAP.0b013e3181e85eb9. PMID 20814282
- [Background] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Background] Persec J, Persec Z, Kopljar M, Zupcic M, Sakic L, Zrinjscak IK, Marinic DK. Low-dose dexamethasone with levobupivacaine improves analgesia after supraclavicular brachial plexus blockade. Int Orthop. 2014 Jan;38(1):101-5. doi: 10.1007/s00264-013-2094-z. Epub 2013 Sep 6. PMID 24173676
- [Background] Kim YJ, Lee GY, Kim DY, Kim CH, Baik HJ, Heo S. Dexamathasone added to levobupivacaine improves postoperative analgesia in ultrasound guided interscalene brachial plexus blockade for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Feb;62(2):130-4. doi: 10.4097/kjae.2012.62.2.130. Epub 2012 Feb 20. PMID 22379567
- [Background] Barrington MJ, Watts SA, Gledhill SR, Thomas RD, Said SA, Snyder GL, Tay VS, Jamrozik K. Preliminary results of the Australasian Regional Anaesthesia Collaboration: a prospective audit of more than 7000 peripheral nerve and plexus blocks for neurologic and other complications. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):534-41. doi: 10.1097/aap.0b013e3181ae72e8. PMID 19916206
- [Background] Barrington MJ, Kluger R. Ultrasound guidance reduces the risk of local anesthetic systemic toxicity following peripheral nerve blockade. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):289-99. doi: 10.1097/AAP.0b013e318292669b. PMID 23788067
- [Background] Compere V, Rey N, Baert O, Ouennich A, Fourdrinier V, Roussignol X, Beccari R, Dureuil B. Major complications after 400 continuous popliteal sciatic nerve blocks for post-operative analgesia. Acta Anaesthesiol Scand. 2009 Mar;53(3):339-45. doi: 10.1111/j.1399-6576.2008.01849.x. PMID 19243320